CLINICAL TRIAL: NCT02691429
Title: Applicability of the Acai Fruit (Euterpe Oleracea) Dye for Chromovitrectomy in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Rafael R. Caiado (Unknown); Casa de Saúde São José (Other); Acácio Alves Souza Lima-Filho (Unknown); Eduardo Novais (Unknown); Emmerson Badaró (Unknown); André Maia (Unknown); Rita Sinigaglia-Coimbra (Unknown); Sung Eun S. Watanabe (Unknown); Eduardo B. Rodrigues (Unknown); Michel Eid Farah (Unknown); Mauricio Maia (Unknown)
Responsible Party: Principal Investigator, Mauricio Maia, MD, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ACAI_2015
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Epiretinal Membrane; Macular Hole; Diabetic Retinopathy
Keywords: Vitreoretinal surgery; euterpe oleracea; chromovitrectomy
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations; Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- acai dye (Euterpe oleracea) 10% (Active Comparator): Twenty-four different retina surgeons will operate one of the 24 selected patients, using the standard vitrectomy technique that employs 4 sclerotomies and a 23-gauge system with accessory illumination. All surgeries will be performed using the acai dye (Euterpe oleracea) in the following concentrations: 10% (n=12) or 25% (n=12).
  Immediately after the procedure, each surgeon will be given an evaluation questionnaire to fill-in
  Interventions: Other: Acai dye 10%
- acai dye (Euterpe oleracea) 25% (Active Comparator): Twenty-four different retina surgeons will operate one of the 24 selected patients, using the standard vitrectomy technique that employs 4 sclerotomies and a 23-gauge system with accessory illumination. All surgeries will be performed using the acai dye (Euterpe oleracea) in the following concentrations: 10% (n=12) or 25% (n=12).
  Immediately after the procedure, each surgeon will be given an evaluation questionnaire to fill-in
  Interventions: Other: Acai dye 10%

INTERVENTIONS:
Other: Acai dye 10% — dye to be used during chromovitrectomy in humans
  Other Names: euterpe oleracea dye

SUMMARY:
Our research group tested the toxicity of different dye concentrations extracted from the acai fruit using a rabbit model. The dye extracted from the acai fruit in concentrations of 10% and 25% was found to be safe for vitreoretinal surgery. This initial research represented the landmark research for testing this alternative vital dye in a clinical research in humans.

The aim of the present clinical trial in humans will be to test the applicability of the acai dye in the identification of the posterior hyaloid and ILM during vitreoretinal surgery in humans.

DETAILED DESCRIPTION:
The purpose of the present clinical trial in humans will be to test the impregnation capacity of the acai dye (10 and 25% concentrations) in the identification of the posterior hyaloid and ILM during vitreoretinal surgery in humans.

Twenty-four patients that seek treatment at the Ophthalmology Department of The Federal University of São Paulo will be selected for this study. Inclusion criteria will be patients diagnosed with epiretinal membrane, macular hole or diabetic retinopathy (with or without vitreal hemorrhages, and/or macular edema, and/or vitreomacular traction). All must be indicated for vitrectomy surgery for the removal of the epiretinal membrane and/or internal limiting membrane.

The present clinical trial was approved by the ethics committee of the Federal University of São Paulo (CEP-UNIFESP). All patients will be invited to sign an Informed Consent Form before participating in the study.

Twenty-four different retina surgeons will operate one of the 24 selected patients, using the standard vitrectomy technique that employs 4 sclerotomies and a 23-gauge system with accessory illumination. All surgeries will be performed using the acai dye (Euterpe oleracea) in the following concentrations: 10% (n=12) or 25% (n=12).

Immediately after the procedure, each surgeon will be given an evaluation questionnaire to fill-in.

All patients will be submitted to the following routine pre-operatory evaluations:

1. Physical and pre-anesthesia evaluations - to be performed by the Anesthesiology Team of the São Paulo Hospital.
2. Complete Ophthalmological Examination - that will include:

   1. Visual Acuity Measurements with best correction for both eyes.
   2. Applaination Tonometry (Goldman Tonometer). For this, one drop of anesthetic solution and one drop of fluorescein were instilled in the eye.
   3. Biomicroscopy
   4. Indirect binocular ophthalmoscopy: under mydriasis that will be obtained before each procedure by topical application of tropicamide and phenylephrine.
   5. Retinography and Angiofluoresceinography (with patient under mydriasis- except when "opacidade de meios")
   6. Optical Coherence Tomography (OCT) of the posterior segment (except when "opacidade de meios")
   7. Multifocal Electroretinogram (except when "opacidade de meios")

The vitrectomy surgery will be performed in all patients of this present study using the 23-gauge technique composed of 4 sclerectomies and vitrectomy without 23-gauge sutures.

During surgery, after vitreous removal, the dye extracted from the acai fruit will be slowly injected using a 23 or 25-gauge silicone cannula connected to a 5ml syringe. The objective of the slow injection of the dye is so that it will deposit over the posterior hyloid/peripheral vitreous due to gravity. At this moment, photographic documentation will be performed.

After the dislocation of the posterior hyloid, the removal of the peripheral vitreous and the excess dye, a MachemerTM (Volk, Germany) macula magnifying lens will be used to improve visualization for the removal of the ILM using an intraocular tweezers. If the ILM is not visible, a second injection with the dye will be performed.

At the end of the surgery, all patients will receive medical prescription of drops with antibiotic and corticoid association during 1 week after the procedure, following vitrectomy post-surgical routine.

A questionnaire with 6 questions (ANNEX 1) will be handed to each surgeon after the end of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with epiretinal membrane, macular hole or proliferative diabetic retinopathy (with or without vitreous hemorrhage).
* Indicated for surgical removal of the epiretinal memebrane (with or without removal of the internal limiting membrane).

Exclusion Criteria:

* - Previous ocular pathology
* Glaucoma
* Any other previous ocular infection that would modify ocular anatomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
ocular inflammation | up to 30 days
  signs of ocular inflammation

SECONDARY OUTCOMES:
intraocular pressure | up to 30 days
  increase of intraocular pressure
complications of the posterior segment | up to 30 days
  macular edema

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Maia, Principal Investigator — Federal University of São Paulo UNIFESP
Locations (1):
- Dept of Ophthalmology - UNIFESP/Hospital São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No